CLINICAL TRIAL: NCT07125326
Title: Intermittent Versus Continuous Bladder Catheterization in Epiduralized Laboring Patients: a Non-blinded Randomized Controlled Trial
Brief Title: How the Method of Bladder Emptying After Epidural Placement in Labor Affects Postpartum Voiding
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Elena Lands, Graduate Medical Fellow, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY24030142
Record Dates: First submitted 2025-08-04; First posted 2025-08-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Urinary Retention; Urinary Tract Infection (Diagnosis); Postpartum Acute Urinary Retention; Postpartum Care; Voiding Dysfunction
Keywords: catheterization; foley; catheter; urinary retention; voiding dysfunction; epidural; labor; bladder catheterization
MeSH Terms: conditions — Urinary Retention; Urinary Tract Infections; Disease | interventions — Intermittent Urethral Catheterization

STUDY DESIGN:
Intervention Model Description: Allocation will be determined based on a previously generated randomization scheme created by the NCI Clinical Trials Randomization Tool.
Who Masked: Investigator, Outcomes Assessor
Masking Description: While the patient, nursing team, and delivery providers will not be blinded to the catheterization method, the provider making the diagnosis of postpartum urinary retention will be blinded to the exposure group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intermittent catheterization (Active Comparator)
  Interventions: Procedure: Intermittent catheterization
- Continuous catheterization (Active Comparator)
  Interventions: Procedure: Continuous catheterization

INTERVENTIONS:
Procedure: Intermittent catheterization — intermittent bladder catheterization every four hours, or shorter intervals if volume exceeds 500mL per expert recommendation
  Arms: Intermittent catheterization
Procedure: Continuous catheterization — One catheter is placed in the bladder until pushing
  Arms: Continuous catheterization

SUMMARY:
At least ten percent of patients have postpartum urinary retention or difficulty urinating after birth, which can cause incontinence and other urinary problems long-term. After getting an epidural placed, patients should be numb in their pelvic region. This numbness makes it difficult to feel the need to urinate, so patients need a urinary catheter placed to empty the bladder. Some patients have one catheter placed throughout their labor and others have a catheter placed to empty the bladder then removed every few hours. The investigators are studying whether placing a catheter once or catheterizing multiple times affects the rate of postpartum urinary problems and infection.

DETAILED DESCRIPTION:
This is a randomized controlled trial to assess the effect of bladder catheterization method during labor with epidural anesthesia on the rate of postpartum urinary retention.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients planning vaginal delivery presenting in labor or for induction of labor
* Age 18 years and older
* Live fetus
* Receive epidural anesthesia

Exclusion Criteria:

* those under 18 years old
* those with stillbirth
* those with baseline overactive bladder symptoms, neurogenic bladder diagnoses, or otherwise using bladder catheterization during pregnancy

Patients will be excluded from UTI analyses if:

* they received antibiotics intrapartum
* had bacteriuria diagnosed by a clean catch specimen showing >100,000 CFU/mL of a single bacterial species, regardless of symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Postpartum urinary retention | Three days postpartum
  Urinary retention defined as overt inability to void at six hours after last bladder emptying postpartum or symptomatic incomplete emptying, or covert retention of >150cc urine in the bladder after voiding Collecting number of participants who experience this

SECONDARY OUTCOMES:
Postpartum urinary tract infection | One week postpartum
  Culture-proven urinary tract infection without pre-existing infection documented on admission for delivery Collecting number of participants who experience this
Patient satisfaction | Immediately postpartum
  Title: Patient satisfaction Minimum rating 1, maximum 5, with 5 corresponding to better outcome Each question will be interpreted alone rather than aggregated
Nurse satisfaction | Immediately postpartum
  Title: Nurse satisfaction Minimum rating 1, maximum 5, with 5 corresponding to better outcome Each question will be interpreted alone rather than aggregated
Voiding function at 2 weeks | 2 weeks postpartum
  Urinary Distress Inventory-6 questionnaire answers, to be analyzed individually (0-4) and also summed, with higher total score indicating worse function from 0 to 24
Voiding function at 6 weeks | 6 weeks postpartum
  Urinary Distress Inventory-6 questionnaire answers, to be analyzed individually (0-4) and also summed, with higher total score indicating worse function from 0 to 24
Voiding function at 6 months | 6 months postpartum
  Urinary Distress Inventory-6 questionnaire answers, to be analyzed individually (0-4) and also summed, with higher total score indicating worse function from 0 to 24
Voiding function at one year | one year postpartum
  Urinary Distress Inventory-6 questionnaire answers, to be analyzed individually (0-4) and also summed, with higher total score indicating worse function from 0 to 24

CONTACTS AND LOCATIONS:
Overall Officials: Anna Binstock, MD, Study Chair — UPMC Magee-Womens Hospital
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No